CLINICAL TRIAL: NCT01325181
Title: Prospective Study on the Efficacy and Safety of Intravitreal Ranibizumab Versus Low-fluence Photodynamic Therapy in the Treatment of Chronic Central Serous Chorioretinopathy
Brief Title: Ranibizumab Versus Low-fluence Photodynamic Therapy in the Treatment of Chronic Central Serous Chorioretinopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jang Won Heo (Other)
Collaborators: Novartis Korea Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jang Won Heo, Associate professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOV001
Record Dates: First submitted 2011-03-25; First posted 2011-03-29 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Central Serous Chorioretinopathy
Keywords: Chronic central serous chorioretinopathy; Ranibizumab; Photodynamic therapy
MeSH Terms: interventions — Verteporfin; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-fluence PDT with Verteporfin (Active Comparator): Half the regular laser fluence PDT(Visudyne®; Novartis); a total light energy of 25J/cm2, a light dose rate of 300mW/cm2. If subretinal fluid was sustained after primary treatment, rescue treatment(ranibizumab injection) was considered
  Interventions: Drug: Verteporfin
- Ranibizumab (Active Comparator): Consecutive Intravitreal injection of ranibizumab(Lucentis®, Novartis) 0.5mg/0.05ml for the first 3 months. If subretinal fluid was sustained after primary treatment, rescue treatment(low-fluence photodynamic therapy) was considered
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: Verteporfin — a 6mg/m2 infusion of verteporfin(Visudyne; Novartis)over 10 minutes followed by laser delivery
  Other Names: Visudyne
  Arms: Low-fluence PDT with Verteporfin
Drug: ranibizumab — Consecutive intravitreal injection of ranibizumab(Lucentis®, Novartis) 0.5mg/0.05ml for the first 3 months
  Other Names: Lucentis
  Arms: Ranibizumab

SUMMARY:
The purpose of this study is to compare the efficacy and safety of intravitreal ranibizumab injection versus low-fluence PDT in the treatment of chronic CSC.

DETAILED DESCRIPTION:
Central serous chorioretinopathy (CSC) is characterized by serous detachment of the neurosensory retina. The pathophysiology of CSC is not certain and various theories are proposed including impaired function of retinal pigment epithelium (RPE), choroidal ischemia and choroidal hyperpermeability leading to RPE damage. Acute CSC with monofocal or paucifocal changes of RPE usually shows spontaneous resolution and has a favorable visual outcome. Chronic CSC is characterized by multifocal or diffuse decompensation of RPE associated with persistent detachment of neurosensory retina. This might lead to cystoid macular degeneration, foveal atrophy and damage to the foveal photoreceptor layer, consequently resulting in irreversible significant visual loss. Photodynamic therapy (PDT) was proposed for the treatment of chronic CSC. Modified parameters of PDT such as shortening of the time of laser emission and reduction of a total light energy have been suggested to reduce the irreversible damages induced by conventional PDT. Recently, intravitreal injection of antibody to vascular endothelial growth factor(VEGF) was proposed as a new treatment option based on the effect of anti-permeability. Several reports demonstrated acceptable outcomes after intravitreal bevacizumab injection, one of anti-VEGF agent. But the clinical results with ranibizumab are not reported yet. The purpose of this study is to compare the efficacy and safety of intravitreal ranibizumab injection versus low-fluence PDT in the treatment of chronic CSC.

ELIGIBILITY:
Inclusion Criteria:

1. best-corrected visual acuity (BCVA) between 0.0 and 1.0 logarithm of the minimal angle of resolution (logMAR)
2. presence of subfoveal fluid persisting for 3 months or more on optical coherence tomography (OCT)
3. presence of leakage and multifocal/diffuse RPE decompensation on fluorescein angiography (FA)
4. choroidal vascular hyperpermeability and abnormal dilation of choroidal vasculature on indocyanine angiography (ICGA)

Exclusion Criteria:

1. previous treatment, such as laser photocoagulation, PDT, intravitreal injection of steroid or anti-VEGF agent
2. evidence of choroidal neovascularization
3. any other ocular diseases that could affect visual acuity
4. systemic steroid treatment in the previous 12 months
5. media opacity such as cataract that could interfere with adequate acquisition of OCT, FA and ICGA images

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jang Won Heo, Professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- • Department of Ophthalmology, Seoul National University College of Medicine, Seoul, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203
- [Derived] Bae SH, Heo JW, Kim C, Kim TW, Lee JY, Song SJ, Park TK, Moon SW, Chung H. A randomized pilot study of low-fluence photodynamic therapy versus intravitreal ranibizumab for chronic central serous chorioretinopathy. Am J Ophthalmol. 2011 Nov;152(5):784-92.e2. doi: 10.1016/j.ajo.2011.04.008. Epub 2011 Jul 13. PMID 21742303

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-fluence PDT | Ranibizumab
Started | 18 | 16
Completed | 18 | 14
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-fluence PDT | Ranibizumab | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 16 | 34
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 51.4 (8.2) | 48.9 (7.5) | 50.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 15 | 13 | 28
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 18 | 16 | 34

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in logMAR BCVA
Description: the changes from baseline in logMAR BCVA throughout the follow-up period
Time Frame: 12 months
Reporting Status: Not Posted

2. Primary Outcome: Number of Participants That Achieved Complete Resolution of Subretinal Fluid on OCT Without Rescue Treatment
Description: number of participants who achieved complete resolution of subretinal fluid on OCT without rescue treatment until the end of the study
Time Frame: 12 months
Population: All study eyes were analyzed using intention to treat principle and the last observation forward method
Measure: Number; unit: participants
Arm/Group | Low-fluence PDT | Ranibizumab
Number analyzed (Participants) | 18 | 16
participants | 16 | 2

3. Secondary Outcome: Change From Baseline in Central Foveal Thickness on OCT
Description: the change from baseline in central foveal thickness measured by OCT throughout the follow-up period
Time Frame: 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Number of Participants With Leakage on Fluorescein Angiography
Description: number of participants who showed fluorescein leakage after primary or rescue treatment throughout the follow-up period
Time Frame: 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Choroidal Hyperpermeability on Indocyanine Green Angiography
Description: change from baseline in the status of choroidal perfusion and hyperpermeability on indocyanine green angiography throughout the follow-up period
Time Frame: 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Number of Participants Who Underwent Rescue Treatment
Description: number of participants who underwent rescue treatment: ranibizumab injections for the low-fluence PDT group and low-fluence PDT for the ranibizumab group
Time Frame: 12 months
Reporting Status: Not Posted

7. Secondary Outcome: Number of Participants With Adverse Event
Description: number of participants with adverse event throughout the follow-up period including procedure and drug-related adverse events
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Low-fluence PDT | Ranibizumab
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No